CLINICAL TRIAL: NCT02566226
Title: Impact of Intrathecal Morphine on Sleep Apnea Syndrome After Hip Arthroplasty Performed Under Spinal Anaesthesia
Brief Title: Impact of Intrathecal Morphine on Sleep Apnea Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Program Director, Regional Anaesthesia, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CER 265/15
Record Dates: First submitted 2015-09-28; First posted 2015-10-02 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine with normal saline (Placebo Comparator)
  Interventions: Drug: Bupivacaine with normal saline
- Bupivacaine with intrathecal morphine (Active Comparator)
  Interventions: Drug: Bupivacaine with intrathecal morphine

INTERVENTIONS:
Drug: Bupivacaine with normal saline — Isobaric bupivacaine 15 mg + normal saline 0.5 cc
  Arms: Bupivacaine with normal saline
Drug: Bupivacaine with intrathecal morphine — Isobaric bupivacaine 15 mg + intrathecal morphine 100 mcg
  Arms: Bupivacaine with intrathecal morphine

SUMMARY:
Intrathecal morphine is commonly used as an analgesic adjunct for hip arthroplasty performed under spinal anaesthesia. Sleep apnea syndrome is a condition that affects up to 10% of the patients. Effect of intrathecal hydrophilic opioids on the frequency and duration of apneic episodes is unknown. The objective of this randomised controlled trial is to investigate the effect of intrathecal morphine and surgery on apneic episodes.

ELIGIBILITY:
Inclusion Criteria:

* physical status I - III
* patients scheduled to undergo hip arthroplasty

Exclusion Criteria:

* planned surgical duration more than 3 hours
* contraindication to spinal anaesthesia
* severe respiratory disease
* patient known and treated for sleep apnea syndrome

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
apnea hypopnea index while lying supine | postoperative night 0

SECONDARY OUTCOMES:
apnea hypopnea index while lying in another position than supine | postoperative night 0
mean pulse oxymetry | postoperative night 0
STOP-BANG questionnaire | 24 h before surgery
Berlin questionnaire | 24 h before surgery
Epworth questionnaire | 24 h before surgery
pain scores (numeric rating scale, 0-10) | postoperative day 0, 1, 2 and 3
oxycodone consumption (mg) | postoperative day 0, 1, 2 and 3
postoperative nausea and vomiting (yes/no) | postoperative day 0, 1, 2 and 3
Pruritus (yes/no) | postoperative day 0, 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Eric Albrecht, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Switzerland

REFERENCES:
- [Derived] Albrecht E, Wegrzyn J, Rossel JB, Bayon V, Heinzer R. Impact of spinal versus general anaesthesia on perioperative obstructive sleep apnoea severity in patients undergoing hip arthroplasty: a post hoc analysis of two randomised controlled trials. Br J Anaesth. 2024 Aug;133(2):416-423. doi: 10.1016/j.bja.2024.04.051. Epub 2024 Jun 10. PMID 38862381
- [Derived] Albrecht E, Bayon V, Hirotsu C, Al Ja'bari A, Heinzer R. Intrathecal morphine and sleep apnoea severity in patients undergoing hip arthroplasty: a randomised, controlled, triple-blinded trial. Br J Anaesth. 2020 Nov;125(5):811-817. doi: 10.1016/j.bja.2020.07.052. Epub 2020 Sep 6. PMID 32900508